CLINICAL TRIAL: NCT01070030
Title: Multi-center, Open Label, 18-week Study to Demonstrate the Efficacy and Safety of Combination Therapy of Aliskiren/Amlodipine or Aliskiren/Amlodipine/Hydrochlorothiazide in Patients With Stage II HT
Brief Title: Efficacy and Safety of Combination Therapy of Aliskiren/Amlodipine or Aliskiren/Amlodipine/Hydrochlorothiazide in Patients With Stage II Hypertension
Acronym: ACADEMY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPP100ATH01
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Stage II Hypertension
Keywords: Stage II Hypertension, Aliskiren, Amlodipine, Hydrochlorothiazide
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Amlodipine

INTERVENTIONS:
Drug: Aliskiren/Amlodipine (150/5 mg/day, 300/10 mg/day) , Aliskiren/Amlodipine/Hydrochlorothiazide (300/10/12.5 mg/day, 300/10/25 mg/day) — The patients were asked for 2 week run-in phase with atenolol 50 mg qd(once a day), followed by 4 schedule visits with 4-week interval until patient achieved BP goal. The maximum follow up was 16-week treatment. At visit 2, the patients started receiving Aliskiren/Amlodipine (150/5mg per day) for 4 weeks. At visit 3, if the patients did not achieve blood pressure (BP) goal, patients were up titrated to Aliskiren/Amlodipine (300/10 mg/day) for 4 weeks. At visit 4, if the patients did not achieve BP goal, HCT 12.5 mg/day was added to Aliskiren/Amlodipine/HCT (300/10/12.5 mg/day) for 4 weeks. Finally at visit 5, if the patients did not achieve BP goal, HCT was up titrated to Aliskiren/Amlodipine/HCT (300/10/25 mg/day) for 4 weeks until visit 6. Once the patients achieved BP goal at any visit, they completed the study.

SUMMARY:
This study assessed the efficacy and safety of combination therapy of Aliskiren/Amlodipine or Aliskiren/Amlodipine/Hydrochlorothiazide in patients with stage II Hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients 18 years of age or older
* Male or female patients are eligible. Female patients must be either post-menopausal for one year, surgically sterile, or using effective contraceptive methods such as oral contraceptives, barrier method with spermicidal or an intrauterine device.
* Patients with a diagnosis of hypertension as following msDBP & msSBP Requirements:

  * For newly diagnosed/untreated patients:

    * Mean Sitting Diastolic Blood Pressure (msDBP) ≥ 100 and < 120 mmHg, and/or mean sitting Systolic Blood Pressure (msSBP) ≥ 160 and < 200 mmHg at Visit1.
  * For previously treated patients with 1 or 2 antihypertensive medications:

    * msDBP ≥ 90 and < 100 mmHg, and/or msSBP ≥ 140 and < 160 mmHg at Visit 1 AND
    * msDBP ≥ 100 and < 120 mmHg, and/or msSBP ≥ 160 and < 200 mmHg at Visit 2.
  * For previously treated patients with Atenolol 50 mg once daily alone more than 2 weeks consecutively at visit 1:

    * msDBP ≥ 100 and < 120 mmHg, and/or msSBP ≥ 160 and < 200 mmHg.
* Patients who are eligible and able to participate in the study, and who consent to do so after the purpose and nature of the investigation has been clearly explained to them (written informed consent).

Exclusion Criteria:

* Patients that previously participated in any Aliskiren study.
* Inability to receive or completely replace all previous antihypertensive medications with Atenolol 50 mg once daily for a period of 2 weeks as required by the protocol.
* Patients on 1 (other than Atenolol 50 mg once daily) or 2 antihypertensive drugs with msDBP ≥ 100 mmHg and/or msSBP ≥ 160 mmHg at Visit 1.
* Patients on 3 or more antihypertensive drugs at Visit 1.
* Pregnant or nursing (lactating) women, when pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (≥ 5 mIU/mL).
* Sexually active female patients who are not using effective contraceptive methods.
* Serum potassium <3.5 mEq/L (mmol/L) or > 5.5 mEq/L at Visit 1.
* Second or third degree heart block with or without a pacemaker, or other potentially life-threatening or symptomatic arrhythmia current or by history.
* History of noncompliance to medical regimens or unwillingness to comply with the study protocol.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with stage II hypertension achieving blood pressure (BP) goal | 18 weeks
  The BP goal for non-diabetic patient is defined as msSBP < 140 mmHg and msDBP < 90 mmHg. The BP goal for diabetic patient is msSBP < 130 mmHg and msDBP < 80 mmHg) in patients with stage II hypertension.

SECONDARY OUTCOMES:
Percentage of participants who have blood pressure surge to their baseline level during 24-h ambulatory blood pressure monitor (ABPM) | 18 weeks
  24-h ABPM profiles were assessed by percentage of participants who have blood pressure (BP) surge to their baseline level (during 24-h ABPM) once after patients achieve BP goal (BP goal for non-diabetic patient is defined as msSBP < 140 mmHg and msDBP < 90 mmHg; and the BP goal for diabetic patient is msSBP < 130 mmHg and msDBP < 80) at any visit only in selected study sites. The mean 24-hour MADBP (Mean Ambulatory Diastolic Blood Pressure) or MASBP (Mean Ambulatory Systolic Blood Pressure) is defined as the average of the hourly MADBP or MASBP over 24 hours respectively.
Change in Mean Sitting Systolic Blood Pressure (msSBP) and Mean Sitting Diastolic Blood Pressure (msDBP) from baseline to study end | From baseline to study completion (between week 8 to 18)
  mSBP and mDBP is defined as an average of 2 points blood pressure measurements which 5 minutes apart. Patient must be at rest for at least 5 minutes in sitting position before the heart rate and blood pressure measurement. The arm for blood pressure measurement should be the same during the whole study.
Number of participants with responder rate for Mean Sitting Systolic Blood Pressure (msSBP) and Mean Sitting Diastolic Blood Pressure (msDBP) | 18 weeks
  The responder rate of msSBP is defined as msSBP < 140 mmHg for non-diabetic patients (msSBP < 130 mmHg for diabetic patients) or by a reduction of ≥ 20 mmHg BP from baseline.
  The responder rate of msDBP is defined as msDBP < 90 mmHg for non-diabetic patients ( msDBP < 80 mmHg for diabetic patients) or by a reduction of ≥ 10 mm Hg BP from baseline
Number of patients with any adverse events | 18 weeks
  An adverse event can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug, whether or not considered related to the medicinal (investigational) product.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Thailand (3):
  - Investigative Site, Bangkok
  - Investigative Site, Chiang Mai
  - Investigative Site, Nakhon Ratchasima